CLINICAL TRIAL: NCT00666549
Title: Research Tissue Bank
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: GCO 07-0548-00106; P01CA108671-01A2 (NIH); MPD-RC 106 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Myelofibrosis; Idiopathic Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera
Keywords: Myeloproliferative Disease; Myelofibrosis; Idiopathic Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, bone marrow, bone marrow biopsy, toenail clippings, phlebotomized blood, spleen cells
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study that will allow for the preservation and/or storage of a small portion one or more of the following tissues:

* Peripheral blood
* Bone marrow
* Bone marrow biopsy
* A phlebotomized unit of blood
* Spleen cells
* Toenail clippings

This material will be used for the study of Myeloproliferative Disorders (MPD) by researchers. The goals of this research study are to understand the causes of MPDs, how to diagnose them more easily and how to treat them better. MPD is a disease affecting hematopoietic stem cells. Hematopoietic stem cells are cells that make blood cells. These stem cells grow in the center portion of the bones called bone marrow. Under some conditions, these cells are also found in blood. There are several diseases, which are classified as MPD. These include polycythemia vera (too many red blood cells), essential thrombocythemia (too many platelets), and idiopathic myelofibrosis (abnormal blood cells and fibers build up in the bone marrow). These syndromes carry a high risk of developing leukemia. It is important to continue to learn more about these blood cancers and to learn more about the effectiveness and potential side effects of various treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Philadelphia chromosome negative myeloproliferative disorders (MPD) polycythemia vera (PV), idiopathic myelofibrosis (IM), and essential thrombocythemia (ET) are eligible.
* Newly diagnose MPD patients as well as previously treated for a MPD are eligible.
* Signed informed consent is required from each patient at the time of enrollment.

Exclusion Criteria:

* Patients currently participating in experimental treatment arms of MPD-RC protocols, or other experimental treatment protocols are not eligible during the period they are on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Philadelphia chromosome negative myeloproliferative disorders (MPD) polycythemia vera (PV), idiopathic myelofibrosis (IM), and essential thrombocythemia (ET) are eligible and not currently participating in any MPD-RC treatment studies.
Sampling Method: Non-Probability Sample
Enrollment: 963 (Actual)
Dates: Start 2007-09; Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

PRIMARY OUTCOMES:
To collect and store tissue specimens from patients with MPDs including PV, IM, ET. The samples will be used to conduct laboratory investigations to help define mechanisms involved in the pathophysiology and treatment of these disorders. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Rona S Weinberg, PhD, Study Chair — Myeloproliferative Disorders-Research Consortium; Lewis Silverman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (11):
- United States (9):
  - Palo Alto Medical Foundation Research Institute, Palo Alto, California
  - Weill Cornell University, Washington D.C., District of Columbia
  - University of Georgetown, Washington D.C., District of Columbia
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Roswell Park, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Italy (2):
  - Ospedali Riuniti di Bergamo, Bergamo, IL
  - University of Florence, Florence, IL